CLINICAL TRIAL: NCT04582227
Title: The Effect of Using Ambu Aura-i Laryngeal Mask Airway Versus Endotracheal Tube on Emergence Hypertension in Supratentorial Cranial Surgery: A Randomized Controlled Study
Brief Title: Using Ambu Aura-i Laryngeal Mask Airway in Cranial Surgery
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Samir Wahdan, Lecturer of Anesthesia, Pain management and Surgical ICU, Cairo University
Other Study IDs: MD-202-2020
Record Dates: First submitted 2020-10-03; First posted 2020-10-09 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Hypertension, Malignant; Airway Management
Keywords: Hypertension; airway; Laryngeal Mask Airway
MeSH Terms: conditions — Hypertension, Malignant; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The ETT group: Oral endotracheal intubation via direct laryngoscopy will be performed. The ETT cuff will be inflated to 25 cmH2O using a manometer.
- The LMA group: The Ambu aura-i LMA size will be chosen and inserted using the recommended single-handed rotational technique. Subsequently, a manometer was used to inflate the cuff to 60 cm H2O.
  Interventions: Device: Ambu aura-i LMA

INTERVENTIONS:
Device: Ambu aura-i LMA — The ETT or the LMA will be inserted with the patient's head position is aided either by pins or head rest, and either the head will be in neutral position or tilted as long as the airway device is successfully placed.
  Groups: The LMA group

SUMMARY:
the investigators hypothesize that Ambu aura-i LMA can be used safely in patients undergoing craniotomies and are effective in reducing the incidence of emergence hypertension.

DETAILED DESCRIPTION:
In this study the investigators want to assess the safety of using SGA devices in cranial surgery and comparing the effect of these devices with ETT regarding hemodynamics stability throughout the procedure and intracranial tension.

ELIGIBILITY:
Inclusion Criteria:

1. Study will be conducted on patients undergoing craniotomies under general anaesthesia in supine position.
2. Aged 18 to 60 years.
3. ASA 1 or 2.
4. GCS ≥ 13.

Exclusion Criteria:

1. Patients who are known hypertensive, history of cardiac diseases or chest diseases
2. Patients with risk of aspiration (Obesity with BMI ≥ 40, hiatal hernia, esophageal cancer and previous esophageal surgery).
3. Risk of difficult intubation
4. Extensive intracranial tumours that may affect recovery of patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients aged from 18 to 60 years presented with brain lesions undergoing craniotomies under general anaesthesia in supine position.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Measure Mean blood pressure | UP TO 1 HOURE
  incidence of emergence hypertension

SECONDARY OUTCOMES:
Measure Mean Heart rate | UP TO 1 HOURE
  incidence of tachycardia or bradycardia with emergence.
successful placement of the airway device | UP TO 1 HOURE
  Number of attempts needed for successful placement of the airway device
incidence of postoperative complication | up to 24 hours
  incidence of postoperative sore throat , hoarseness
amount of fentanyl | up to 24 hours
  by microgram

CONTACTS AND LOCATIONS:
Overall Officials: Amr s wahdan, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided